CLINICAL TRIAL: NCT03803345
Title: The Association of Maternal Night-Eating Pattern With Glucose Tolerance During Pregnancy
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University of Singapore (Other); National University Hospital, Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB 2018/2529
Record Dates: First submitted 2018-12-18; First posted 2019-01-14 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Metabolic Disease
Keywords: Food timing; Gestational diabetes mellitus; Glucose tolerance; Night-eating; Pregnancy outcomes; Snacking
MeSH Terms: conditions — Metabolic Diseases; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the associations of maternal food timing with glucose levels during pregnancy.

DETAILED DESCRIPTION:
A novel line of research has emerged, suggesting that synchronizing the timing of food intake with body's circadian rhythms or day-night cycle has metabolic implications. Eating at the inappropriate time can disrupt circadian system which might induce metabolic perturbations, including glucose abnormalities. Recent evidence showed that circadian timing of eating was associated with glucose regulation in pregnant women. However, little is known about night-eating pattern during pregnancy, particularly the influence of nocturnal snacking on glycaemic control.

This cross-sectional study aims to recruit 400 pregnant women at 18-21 weeks' gestation. The investigators will assess maternal dietary intake, monitor 24-hour activity-rest pattern and light-dark exposure, and measure glucose and insulin profiles during the second trimester of pregnancy. Maternal socio-demographic status, lifestyle characteristics, health conditions and pregnancy outcomes will be asked through interview or retrieved from medical notes.

This study allows understanding the importance of circadian eating pattern, which is a modifiable behavior, in glycaemic control during pregnancy, and help to provide evidence for developing nutritional guidelines which can ameliorate metabolic health for mothers.

ELIGIBILITY:
Inclusion Criteria:

1. 18-21 week's gestation
2. Singapore citizens or Singapore Permanent Residents
3. Age 18-45 years
4. Plan to follow-up for antenatal care in KK Women's and Children's Hospital
5. Intend to deliver in KK Women's and Children's Hospital
6. Provide written informed consent

Exclusion Criteria:

1. Type 1 or 2 diabetes
2. Diabetes in pregnancy as confirmed by oral glucose tolerance test
3. Use of medications such as anticonvulsant medications or oral steroids in the past 1 month
4. Multiple pregnancy
5. On routine night-shift work for at least 3x/week over the past 1 month
6. Known or suspected allergy to medical grade adhesives
7. Chronic kidney diseases
8. Preeclampsia
9. Eventual miscarriage or undergo termination event

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women.
Study Population: Healthy pregnant women aged 18-45 years old and at 18-21 weeks of gestation upon recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Maternal glucose tolerance | Up to 4 weeks, during second trimester of pregnancy
  Maternal glucose tolerance based on plasma glucose levels as assessed by the Oral Glucose Tolerance Test.
Maternal night-eating pattern | Up to 4 days, during second trimester of pregnancy
  Maternal night-eating pattern as assessed by the food diary and food record app.
Maternal meal and snack distribution | Up to 4 days, during second trimester of pregnancy
  Maternal meal and snack distribution as assessed by the food diary and food record app.

SECONDARY OUTCOMES:
Maternal insulin profile | Up to 4 weeks, during second trimester of pregnancy
  Maternal insulin profile as assessed by the fasting insulin level.
Maternal gestational diabetes status | up to 4 weeks, during second trimester of pregnancy
  Maternal gestational diabetes status as assessed by the Oral Glucose Tolerance Test.
Maternal glycemic variability | Up to 10 days, during second trimester of pregnancy
  Maternal glycemic variability based on continuous glucose monitoring profile as assessed by the continuous glucose monitoring system (Freestyle Libre Pro, Abbott).
Maternal diet quality | up to 1 month, during second trimester of pregnancy
  Maternal diet quality as assessed by the Food Frequency Questionnaire.
Maternal type of food intake | up to 10 weeks, during second trimester of pregnancy
  Maternal type of food intake as assessed by the food diary, food record app and Food Frequency Questionnaire.
Maternal nutritional intake | Up to 4 days, during second trimester of pregnancy
  Maternal nutritional intake as assessed by the food diary and food record app.
Maternal eating frequency | Up to 4 days, during second trimester of pregnancy
  Maternal eating frequency as assessed by the food diary and food record app.
Maternal meal and snack regularity | Up to 1 month, during second trimester of pregnancy
  Maternal meal and snack regularity as assessed by the questionnaire based on frequency of meal/ snack delay and skipping.
Maternal physical activity | Up to 10 days, during second trimester of pregnancy
  Maternal physical activity as measured by the Actigraph accelerometer.
Maternal physical activity | Up to 1 week, during second trimester of pregnancy
  Maternal physical activity as assessed using the modified International Physical Activity Questionnaire (IPAQ).
Maternal sedentary behavior | Up to 10 days, during second trimester of pregnancy
  Maternal sedentary behavior as measured by the Actigraph accelerometer.
Maternal sedentary behavior | Up to 1 week, during second trimester of pregnancy
  Maternal sedentary behavior as assessed using the structured questionnaires based on frequency and duration of time spent in sedentary behaviour.
Maternal sleep related behavior | Up to 10 days, during second trimester of pregnancy
  Maternal sleep related behaviour as measured by the Actigraph accelerometer.
Maternal sleep related behavior | Up to 1 month, during second trimester of pregnancy
  Maternal sleep related behavior as assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire.
Maternal light exposure | Up to 10 days, during second trimester of pregnancy
  Maternal light exposure as measured by the Actigraph accelerometer.
Maternal light exposure | Up to 1 week, during second trimester of pregnancy
  Maternal light exposure as assessed by the Harvard Light Exposure Assessment (H-LEA) questionnaire.
Maternal electronic media use before bedtime | up to 1 week, during second trimester of pregnancy
  Maternal electronic media use before bedtime as assessed by the structured questionnaire based on frequency, duration and location of electronic device use.
Maternal mood | Up to 1 week, during second trimester of pregnancy
  Maternal mood as assessed by the Depression Anxiety Stress Scale (DASS21) questionnaire.
Maternal gestational weight gain | Up to 42 weeks, throughout pregnancy
  Maternal weight measured by calibrated weighing scale as recorded in medical notes
Dietary data from food record app. | up to 4 days, during second trimester of pregnancy
  Feasibility and validity of using food record mobile app to capture maternal dietary intake, compared with paper-based food diary.

OTHER OUTCOMES:
Maternal hypertension status | Up to 42 weeks, during pregnancy
  Maternal hypertension status obtained from medical notes.
Maternal delivery outcomes | Up to 72 hours, after delivery
  Maternal delivery outcomes obtained from medical notes.
Birth weight | Up to 72 hours, after delivery
  Offspring birth weight in gram obtained from medical notes.
Birth length | Up to 72 hours, after delivery
  Offspring birth length in cm obtained from medical notes.
Birth head circumference | Up to 72 hours, after delivery
  Offspring birth head circumference in cm obtained from medical notes.

CONTACTS AND LOCATIONS:
Overall Officials: See Ling Loy, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YE, Ku CW, Chong MF, Yap F, Chan JKY, Loy SL, Chen LW. Associations of >1-h compared with 1-h meal timing variability (eating jetlag) with plasma glycemic parameters and continuous glucose monitoring measures among pregnant females: a prospective cohort study. Am J Clin Nutr. 2025 Jul;122(1):244-254. doi: 10.1016/j.ajcnut.2025.04.026. Epub 2025 Apr 26. PMID 40294750
- [Derived] Loy SL, Cheung YB, Chong M, Muller-Riemenschneider F, Lek N, Lee YS, Tan KH, Chern B, Yap F, Chan J. Maternal night-eating pattern and glucose tolerance during pregnancy: study protocol for a longitudinal study. BMJ Open. 2019 Oct 10;9(10):e030036. doi: 10.1136/bmjopen-2019-030036. PMID 31601588